CLINICAL TRIAL: NCT05897437
Title: Investigating the Fine and Gross Motor Performance in Children With Attention Deficit Hyperactivity Disorder
Brief Title: Motor Performance in Children With Attention Deficit Hyperactivity Disorder
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ozgun Kaya Kara, Assoc. Prof. PhD, Akdeniz University
Other Study IDs: 2020-271
Record Dates: First submitted 2023-06-01; First posted 2023-06-09 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-07

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: attention deficit hyperactivity disorder; motor skills; Children
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ADHD group: Children with ADHD
- Control Group: Typically developing children

SUMMARY:
Attention deficit hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders in children. Children with ADHD have difficulties with co-contraction, producing muscle force, and regulating movement velocity, and physical fitness. The purpose of this study was to compare the gross and fine motor abilities in children with ADHD and children with typical development.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD) is one of the most common neurodevelopmental disorders in children worldwide with a prevalence of 2.6-4.5% between the ages of 6 and 18 years. When compared to children with typical development, children with ADHD have lower scores in 9-12% of gross motor abilities, 9-36% of balance and postural control, 9-19% of fine motor abilities, and 19-22 % of manual and body coordination. Furthermore, children with ADHD have difficulties with co-contraction, producing muscle force, and regulating movement velocity, and physical fitness. As a consequence of the core symptoms of ADHD, such as inattention, impulsivity, and hyperactivity, over 30-50% of children with ADHD may have impaired motor ability. The purpose of this study was to compare the gross and fine motor abilities in children with ADHD and children with typical development.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of children with attention deficit hyperactivity disorder
* aged at 6 -15 years old
* able to understand and accept verbal instructions.

Exclusion Criteria:

* Clinical diagnosis of children with another psychiatric including autism spectrum disorder, psychotic symptoms, depression
* Clinical diagnosis of children with neurological disorder including cerebral palsy, epilepsy, or speech impairments
* the parents declined to participate in the study.

Ages: 6 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The children with ADHD
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2023-09-03 (Estimated); Study Completion 2023-09-16 (Estimated)

PRIMARY OUTCOMES:
Motor Proficiency | One day
  The Bruininks-Oseretsky Motor Proficiency Test-2 (BOT-2) was used for the evaluation of gross and fine motor skills

CONTACTS AND LOCATIONS:
Overall Officials: Ozgun Kaya Kara, Assoc. Prof., Principal Investigator — Akdeniz University
Locations (1):
- Akdeniz University, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Polanczyk GV, Salum GA, Sugaya LS, Caye A, Rohde LA. Annual research review: A meta-analysis of the worldwide prevalence of mental disorders in children and adolescents. J Child Psychol Psychiatry. 2015 Mar;56(3):345-65. doi: 10.1111/jcpp.12381. Epub 2015 Feb 3. PMID 25649325
- [Background] Goulardins JB, Marques JC, Casella EB, Nascimento RO, Oliveira JA. Motor profile of children with attention deficit hyperactivity disorder, combined type. Res Dev Disabil. 2013 Jan;34(1):40-5. doi: 10.1016/j.ridd.2012.07.014. Epub 2012 Aug 30. PMID 22940157
- [Background] Cho H, Ji S, Chung S, Kim M, Joung YS. Motor function in school-aged children with attention-deficit/hyperactivity disorder in Korea. Psychiatry Investig. 2014 Jul;11(3):223-7. doi: 10.4306/pi.2014.11.3.223. Epub 2014 Jul 21. PMID 25110492
- [Background] Mao HY, Kuo LC, Yang AL, Su CT. Balance in children with attention deficit hyperactivity disorder-combined type. Res Dev Disabil. 2014 Jun;35(6):1252-8. doi: 10.1016/j.ridd.2014.03.020. Epub 2014 Mar 28. PMID 24685941
- [Background] Rosa Neto F, Goulardins JB, Rigoli D, Piek JP, Oliveira JA. Motor development of children with attention deficit hyperactivity disorder. Braz J Psychiatry. 2015 Jul-Sep;37(3):228-34. doi: 10.1590/1516-4446-2014-1533. PMID 26376053